CLINICAL TRIAL: NCT00440479
Title: An Observational Study To Determine Velcade (Bortezomib) Safety and Effectiveness at First Relapse After Participation In First Line HOVON-49/50 Clinical Studies (ADVANCE)
Brief Title: ADVANCE: An Observational Study To Determine Bortezomib Safety and Effectiveness at First Relapse After Participation In First Line HOVON-49/50 Clinical Studies.
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012361; 26866138MMY4013
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma; Hematological Neoplasms
Keywords: Multiple Myeloma; hematological neoplasms; chemotherapy; efficacy; safety; bortezomib; proteasome inhibitor
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Bortezomib dose as determined (observational study) by treating physician
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — dose as determined (observational study) by treating physician

SUMMARY:
The primary aim of this observational study is to collect safety and effectiveness data for bortezomib used at first relapse in a group of multiple myeloma patients who received specific and well defined first line treatments within previous clinical studies.

DETAILED DESCRIPTION:
There is a need by physicians to evaluate the results of bortezomib treatment in a homogenous patient population with regard to the multiple myeloma treatments in first line. For that reason the current study, ADVANCE, is designed to structurally collect data on the daily practice use of bortezomib as treatment after first relapse in patients with specific and well defined first line treatments (i.e. patients who participated in the HOVON-49 or HOVON-50 study). In both HOVON studies patients were randomized to either receiving thalidomide or not, as a part of the first line treatment. Therefore, the effect of pre-treatment with thalidomide on duration, effectiveness and safety of the bortezomib treatment after first relapse can be studied specifically. The analysis of this particular type of data will, however, be descriptive. All adverse events, regardless of seriousness, severity, or presumed relationship to bortezomib therapy will be recorded on the case report form, i.e., a form for each patient in the study on which all needed data are recorded, and reported to the sponsor within current timelines. The sponsor assumes responsibility for appropriate reporting of adverse events to the regulatory authorities. This project is a 'post authorization study (PAS)'. This means that only routinely available medical data are collected, with the patients' permission, and no additional interventions or diagnostic procedures should be done specifically for this study. Because the study is observational, dosage, administration and duration of treatment is at discretion of the treating physician

ELIGIBILITY:
Inclusion Criteria:

* Patients have to sign a statement that they agree with collection of their clinical data for this project
* patients had a first relapse or progressive disease after treatment in the HOVON-49 or HOVON-50 study and will be treated with bortezomib.

Exclusion Criteria:

* Prior enrollment in HOVON-54 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients treated with bortezomib at first relapse after participation in first line HOVON 49 or 50 clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2006-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Response to treatment | No timepoints have been defined, as this is an observational study; data will be collected until three years after latest bortezomib administration

SECONDARY OUTCOMES:
bortezomib treatment schedule, dosing and timing | each cycle
combination therapies for multiple myeloma | from start of bortezomib treatment up to 30 days after last bortezomib administration
adverse events | from start of bortezomib treatment up to 30 days after last bortezomib administration
overall survival | from end of bortezomib treatment up to 3 years after last bortezomib administration

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.
Locations (9):
- Netherlands (9):
  - Bergen op Zoom
  - Breda
  - Ede Gld
  - Flushing
  - Nijmegen
  - Rotterdam
  - Terneuzen
  - Tilburg
  - Utrecht